CLINICAL TRIAL: NCT04885010
Title: Probiotics for Athlete's Recovery and Immune System
Brief Title: Probiotics and Overreaching Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PARIS
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Fatigue; Muscle, Heart; Immunosuppression
MeSH Terms: conditions — Fatigue | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): participants will train for 15 days while consuming the dietary supplement. During the last 8 days the intensity of training will increase to induce overreaching.
  Interventions: Dietary Supplement: probiotics
- Placebo (Placebo Comparator): participants will train for 15 days while consuming the dietary supplement. During the last 8 days the intensity of training will increase to induce overreaching.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotics — participants will be given probiotics twice a day for 15 days
  Arms: Probiotics
Dietary Supplement: placebo — participants will be given a placebo twice a day for 15 days
  Arms: Placebo

SUMMARY:
Overloading is a key training principle used by athletes and coaches to improve physical performance. Intensified training periods are therefore commonly incorporated into the course of a regular training season. From a clinical point of view, very intense periods of training are associated with a temporary immunological deficiency which can lead to teh "overreaching syndroms".

During periods of overreaching, nutritional strategies are mainly aimed at ensuring sufficient amounts of energy to support the increase in effort. However less is known about nutritional supplements to attenuated the inflammatory/immunological response to training stress.

Probiotic bacteria are defined as live food ingredients beneficial to the host's health. Numerous health benefits have been attributed to probiotics, including effects on gastrointestinal tract function and disease, immune function, hyperlipidemia, hypertension, and allergic conditions. Studies in the literature on the ergogenic effect of probiotics in athletes are still scarce today. this study aims to explore the potential role of probiotics on performance, recovery from fatigue and immune function during intensive period of training.

ELIGIBILITY:
Inclusion Criteria:

* age 25-55 years
* Body mass index:> 18 and <30 kg / m2
* Stable body weight for at least 3 months
* regular practice of physical activity for at least 2 years

Exclusion Criteria:

* Chronic diseases (cardiovascular, hepatic, respiratory, cancer)
* Acute inflammatory states, infections or other pathologies
* Regular use of probiotics
* Use or treatment with steroids (within the previous 3 months)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
lymphocyte subpopulation total T (CD3+) | Change from baseline to up to 15 days
  lymphocyte subpopulation: total T (CD3+) %
T-helper (CD4+) | Change from baseline to up to 15 days
  lymphocyte subpopulation: T-helper (CD4+) %
T-suppressor (CD8+) | Change from baseline to up to 15 days
  lymphocyte subpopulation: T-suppressor (CD8+) %

IPD SHARING:
Plan to Share IPD: No